CLINICAL TRIAL: NCT01646125
Title: A Multicenter, Open-label, Randomized Phase II Study to Evaluate the Efficacy of AUY922 vs Pemetrexed or Docetaxel in NSCLC Patients With EGFR Mutations Who Have Progressed on Prior EGFR TKI Treatment
Brief Title: An Open-label, Randomized Phase II Study to Evaluate the Efficacy of AUY922 vs Pemetrexed or Docetaxel in NSCLC Patients With EGFR Mutations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: An interim analysis was conducted in May-2014. Upon review of the data, the committee recommended study termination due to futility.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAUY922A2207; 2012-001050-25 (EudraCT Number)
Record Dates: First submitted 2012-06-26; First posted 2012-07-20 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Advanced Non Small Cell Lung Cancer (NSCLC)
Keywords: Non-small cell lung carcinoma (NSCLC); treatment of lung cancer after first metastasis; lung cancer; lung adenocarcinoma; Squamous cell lung carcinoma; Large-cell lung carcinoma; Non small cell lung carcinoma; Non small cell lung cancer; Non-small cell lung cancer; NSCLC; Large cell lung carcinoma; Large cell lung cancer; HSP90; AUY922; Pemetrexed; Docetaxel; EGFR TKI; EGFR mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide; Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AUY922 arm (Experimental): Participants were assigned to one of two treatment arms in a ratio of 1:1. This was the investigational drug arm.
  AUY922 was to be administered weekly.
  Interventions: Drug: AUY922
- chemotherapy arm (Active Comparator): Participants were assigned to one of two treatment arms in a ratio of 1:1. This was the control arm drug arm.
  Pemetrexed or docetaxel was to be was to be given once every three weeks.
  Interventions: Drug: Docetaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: AUY922 — AUY922 was to be given by i.v. once weekly at 70 mg/m2 until disease progression, death or any other reason for discontinuation from study treatment.
  Arms: AUY922 arm
Drug: Docetaxel — Docetaxel was to be given i.v. once every 3 weeks at 75 mg/m2 until progression or unacceptable toxicity
  Other Names: TAXOTERE
  Arms: chemotherapy arm
Drug: Pemetrexed — Pemetrexed was to be given once every 3 weeks at 500 mg/m2 until progression or unacceptable toxicity
  Other Names: ALIMTA
  Arms: chemotherapy arm

SUMMARY:
The purpose of this study was to determine if AUY922 had superior efficacy when compared to chemotherapy agents docetaxel or pemetrexed in patients whose tumor had EGFR mutations.

The primary purpose of this study was to compare the efficacy of AUY922, when administered i.v. on a once-weekly schedule at 70 mg/m2, versus docetaxel or pemetrexed in adult patients with advanced NSCLC, whose tumors harbored EGFR activating mutations, and had developed resistance to EGFR TKI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically documented, locally advanced (stage IIIB who are not amenable to combined modality treatment) or recurrent or metastatic (Stage IV) non-small cell lung cancer.
2. Patients must have EGFR gene mutation in their tumors. This can be source - documented by one of the following:

   • Provide a pathology report that indicates the patient's tumor had EGFR activating mutation in the past.

   Or:

   • Perform testing (local or central) in an archival tumor or a fresh baseline biopsy tumor tissue to show the presence of EGFR activating mutation.
3. Patients must have documented clinical benefit (CR, PR, or patients with SD for 6 months or greater) on prior EGFR TKI (e.g. erlotinib or gefitinib) followed by documented progression according to RECIST.
4. Patients must have received prior platinum containing treatment.
5. WHO performance status of 0-1

Exclusion Criteria:

1. Patients who have received more than two prior lines of antineoplastic therapy for advanced disease. Chemotherapy administered as neoadjuvant or adjuvant treatment more than six months prior to study enrollment is not considered a prior line of therapy for purposes of this study.
2. Evidence of spinal cord compression or current evidence of CNS metastases. Screening CT/MRI of the brain is mandatory. Note: Patients who have been treated for CNS metastases by radiation or gamma knife surgery, who been stable for at least 2 months and have discontinued high dose corticosteroids will be eligible for protocol participation
3. Prior treatment with an HSP90 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-11-23 (Actual); Primary Completion 2015-11-04 (Actual); Study Completion 2015-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- United States (3):
  - Cedars Sinai Medical Center Dept.of Cedars-Sinai Med. Ctr., Los Angeles, California
  - Maryland Oncology Hematology, P.A. SC, Rockville, Maryland
  - University of Wisconsin / Paul P. Carbone Comp Cancer Center Univ Wisc 5, Madison, Wisconsin
- France (3):
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (4):
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Orbassano, TO
- Novartis Investigative Site, Koto Ku, Tokyo, Japan
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
- Novartis Investigative Site, Gdansk, Poland
- South Korea (3):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Taiwan (3):
  - Novartis Investigative Site, Kuei-Shan Chiang, Taoyuan/ Taiwan ROC
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Leicester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized in a ratio of 1:1 to receive either AUY922 or pemetrexed/docetaxel. A total of 59 participants were randomized in the study: 31 to the AUY922 arm and 28 to the chemotherapy arm. 2 patients from the AUY922 arm & 5 from the chemotherapy arm were not treated. Only 52 received at least 1 dose of study medication.
Period: Overall Study
Arm/Group | AUY922 Arm | Chemotherapy Arm
Started | 31 | 28
Completed | 0 | 0
Not Completed | 31 | 28
Not completed — Untreated | 2 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Death | 1 | 1
Not completed — Physician Decision | 1 | 3
Not completed — Progressive disease | 22 | 16
Not completed — Study terminated by sponsor | 2 | 1
Not completed — Subject/Guardian decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) comprised of all patients who were randomized to a study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | AUY922 Arm | Chemotherapy Arm | Total
Number analyzed (Participants) | 31 | 28 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (10.10) | 62.1 (10.34) | 61.9 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 48
  Male | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Compared PFS between the treatment of AUY922 to comparators Pemetrexed or Docetaxel. Progression-free survival (PFS) based on local investigator assessment per RECIST 1.1 was the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient had not had an event, progression-free survival is censored at the date of last adequate tumor assessment. Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 16 months
Population: Efficacy analysis set (EAS) compromised of a subset of patients in the FAS who received 2 lines of prior antineoplastic therapy consisting of a platinum-based treatment & an EGFR TKI treatment. The DMC recommendation at Interim analysis was to stop the study for futility. As a result, collection of all efficacy assessments was stopped.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | AUY922 Arm | Chemotherapy Arm
Number analyzed (Participants) | 19 | 17
Months | 1.5 [1.2 to 5.6] | 2.3 [1.2 to 4.0]
Statistical Analysis 1: Comparison: AUY922 Arm vs Chemotherapy Arm; Test type: Superiority or Other; Cox Proportional Hazard = 0.76, 90% CI 2-sided [0.35 to 1.63]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was to be compared between treatment arms. The ORR was to be based on local investigator assessment per Response Evaluation Criteria In Solid Tumors Criteria 1.1 (RECIST 1.1). Per this criteria for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.This outcome measure was originally planned to be analyzed up to 24 months. The DMC recommendation at the IA was to stop the study for futility. As a result, collection of all the efficacy assessments was stopped at that time.
Time Frame: 16 months
Population: The data monitoring committee's (DMC's) recommendation based on the Interim Analysis (IA) results was to terminate the study early due to futility; collection of efficacy data for assessment was stopped at that time.
Measure: Number; unit: Participants
Arm/Group | AUY922 Arm | Chemotherapy Arm
Number analyzed (Participants) | 19 | 17
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 3 | 2
  ORR (CR + PR) | 3 | 2

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to date of death due to any cause. If a death has not been observed by the date of analysis cutoff, then OS was to be censored at the last known date patient was alive.
Time Frame: from randomization until death up to death
Population: The data monitoring committee (DMC's) recommendation based on the Interim Analysis (IA) results was to terminate the study early due to futility; collection of efficacy data for assessment was stopped at that time.
Arm/Group | AUY922 Arm | Chemotherapy Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Duration of DCR will be compared between treatment arms. The duration of DCR will be based on local investigator assessment per RECIST 1.1
Time Frame: baseline, until disease progression up to 24 months
Population: as for outcome 3
Arm/Group | AUY922 Arm | Chemotherapy Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Response (TRR)
Description: TTR was to compare between treatment arms. The TTR was to be based on local investigator assessment per RECIST 1.1
Time Frame: baseline, until disease progression up to 24 months
Population: as for outcome 3
Arm/Group | AUY922 Arm | Chemotherapy Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of Response (DOR)
Description: The DOR will be compared between treatment arms. The DOR will be based on local investigator assessment per RECIST 1.1
Time Frame: baseline, until disease progression up to 24 months
Population: as for outcome 3
Arm/Group | AUY922 Arm | Chemotherapy Arm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Rate of Adverse Events (AEs)
Description: To evaluate safety and tolerability of AUY922 compared to chemotherapy agents pemetrexed or docetaxel.
Time Frame: baseline, until disease progression up to 24 months
Population: as for outcome 3
Arm/Group | AUY922 Arm | Chemotherapy Arm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Laboratory Paramenters
Description: Changes in hematology and chemistry values, vital signs, electrocardiograms (ECGs), Dose interruptions, reductions and dose intensity.
Time Frame: baseline, until disease progression up to 24 months
Population: as for outcome 3
Arm/Group | AUY922 Arm | Chemotherapy Arm
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Progression (TTP)
Description: TTP will be compared between treatment arms. The TTP will be based on local investigator assessment per RECIST 1.1
Time Frame: baseline, until disease progression up to 24 months
Population: as for outcome 3
Arm/Group | AUY922 Arm | Chemotherapy Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Safety set: comprised of all participants who received at least one dose of study medication (AUY922, pemetrexed or docetaxel). In the safety set, patients were classified and analyzed according to the treatment received. Of the 59 participants randomized, only 52 received one dose of study medication.
Groups:
- Total: Total
Arm/Group | AUY922 Arm | Chemotherapy Arm | Total
Serious Adverse Events (participants affected / at risk) | 10/29 | 6/23 | 16/52
Other Adverse Events (participants affected / at risk) | 28/29 | 21/23 | 49/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AUY922 Arm (N=29) | Chemotherapy Arm (N=23) | Total (N=52)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 1
RETINAL DEGENERATION (Eye disorders) | 1 | 0 | 1
VISION BLURRED (Eye disorders) | 1 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 1
ASTHENIA (General disorders) | 0 | 1 | 1
DISCOMFORT (General disorders) | 1 | 0 | 1
PYREXIA (General disorders) | 0 | 1 | 1
SUDDEN DEATH (General disorders) | 1 | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 1 | 1
PNEUMONIA (Infections and infestations) | 1 | 1 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 1
EPILEPSY (Nervous system disorders) | 1 | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AUY922 Arm (N=29) | Chemotherapy Arm (N=23) | Total (N=52)
ANAEMIA (Blood and lymphatic system disorders) | 5 | 0 | 5
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 | 1 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 3 | 3
ACCOMMODATION DISORDER (Eye disorders) | 2 | 0 | 2
NIGHT BLINDNESS (Eye disorders) | 2 | 0 | 2
PHOTOPSIA (Eye disorders) | 10 | 0 | 10
VISION BLURRED (Eye disorders) | 6 | 0 | 6
VISUAL ACUITY REDUCED (Eye disorders) | 2 | 0 | 2
VISUAL IMPAIRMENT (Eye disorders) | 6 | 0 | 6
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 1 | 3
CONSTIPATION (Gastrointestinal disorders) | 6 | 2 | 8
DIARRHOEA (Gastrointestinal disorders) | 21 | 1 | 22
DRY MOUTH (Gastrointestinal disorders) | 1 | 2 | 3
NAUSEA (Gastrointestinal disorders) | 10 | 3 | 13
STOMATITIS (Gastrointestinal disorders) | 1 | 3 | 4
VOMITING (Gastrointestinal disorders) | 3 | 3 | 6
ASTHENIA (General disorders) | 8 | 8 | 16
AXILLARY PAIN (General disorders) | 2 | 0 | 2
FATIGUE (General disorders) | 10 | 5 | 15
NON-CARDIAC CHEST PAIN (General disorders) | 2 | 1 | 3
OEDEMA PERIPHERAL (General disorders) | 1 | 2 | 3
PYREXIA (General disorders) | 2 | 4 | 6
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 2 | 0 | 2
CONJUNCTIVITIS (Infections and infestations) | 0 | 3 | 3
RHINITIS (Infections and infestations) | 2 | 0 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 1 | 4
URINARY TRACT INFECTION (Infections and infestations) | 1 | 2 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0 | 2
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 | 0 | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 | 3 | 7
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 0 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 0 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 3 | 8
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 | 0 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
DIZZINESS (Nervous system disorders) | 2 | 0 | 2
HEADACHE (Nervous system disorders) | 9 | 0 | 9
PARAESTHESIA (Nervous system disorders) | 2 | 2 | 4
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 | 2 | 4
VISUAL FIELD DEFECT (Nervous system disorders) | 2 | 0 | 2
VISUAL PERSEVERATION (Nervous system disorders) | 2 | 0 | 2
DEPRESSION (Psychiatric disorders) | 2 | 0 | 2
INSOMNIA (Psychiatric disorders) | 3 | 0 | 3
POLLAKIURIA (Renal and urinary disorders) | 2 | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 9
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 9
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 6 | 6
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 6 | 2 | 8
RASH (Skin and subcutaneous tissue disorders) | 2 | 4 | 6
HYPERTENSION (Vascular disorders) | 5 | 0 | 5

LIMITATIONS AND CAVEATS:
The data monitoring committee (DMC's) recommendation based on the Interim Analysis (IA) results to terminate the study early due to futility, data was not collected for this assessment on many of the secondary endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.